CLINICAL TRIAL: NCT04600180
Title: Deep Phenotyping of the Gut Immune System During Immune Checkpoint Inhibitor Therapy - DEFENCE
Brief Title: The Gut Immune System During Immune Checkpoint Inhibitor Therapy
Acronym: DEFENCE
Status: Active, not recruiting | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: 202000666
Record Dates: First submitted 2020-10-19; First posted 2020-10-23 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Cancer
Keywords: Immune Checkpoint Inhibitor; Cancer; Gut Wall
MeSH Terms: conditions — Neoplasms | interventions — Sigmoidoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Gut wall biopsies and venous blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Palliative treatment with immunotherapy
  Interventions: Procedure: sigmoidoscopies and and venous blood sampling

INTERVENTIONS:
Procedure: sigmoidoscopies and and venous blood sampling — Sigmoidoscopies will be performed at baseline and during immunotherapy. During these procedures biopsies will be taken from the sigmoid and rectum. At the same timepoints, venous blood samples will be taken.

SUMMARY:
This exploratory study aims to gain insight in gut immune system phenotypes before and after immunotherapy. After informed consent is obtained, sigmoidoscopies at baseline and during treatment with immunotherapy will be performed, During the endoscopies, biopsies from the sigmoid and rectum will be obtained. Subsequent immune cell analyses in these biopsies will be performed. Parallel to the sigmoidoscopies, venous blood samples will be obtained to monitor inflammatory markers.

ELIGIBILITY:
Inclusion Criteria:

* Indication for treatment with anti PD1/PDL1 based immunotherapy
* Written informed consent
* Evaluable according to iRECIST v1.1

Exclusion Criteria:

* Concomitant, chronic or infectious illness in the past 6 months causing moderate to severe colitis
* Use of a medication in the past 6 months with an elevated risk of moderate to severe colitis
* Gastrointestinal resection or enterostomy
* Abdominal radiotherapy in the past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with cancer and an indication for palliative treatment with immune checkpoint inhibitors.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Estimated)
Dates: Start 2021-10-30 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
CD8+ T cell count in the gut mucosa | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jacco J. de Haan, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided